CLINICAL TRIAL: NCT03689192
Title: Arginase-1 Peptide Vaccine in Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Inge Marie Svane, MD, Professor, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA1809
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Non Small Cell Lung Cancer; Urothelial Carcinoma; Malignant Melanoma; Ovarian Cancer; Colorectal Cancer; Breast Cancer; Squamous Cell Carcinoma of the Head and Neck; Metastatic Cancer
Keywords: Arginase 1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Melanoma; Ovarian Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARG1-18,19,20 peptide vaccine (Experimental): One ARG1-vaccine every third week for 45 weeks.
  Interventions: Biological: ARG1-18,19,20

INTERVENTIONS:
Biological: ARG1-18,19,20 — 300 ug ARG1-18,19,20 peptide in water mixed with 500ul montanide

SUMMARY:
In this phase I first-in-humans-study a vaccine consisting of arginase-1 (ARG1) peptides and the adjuvant Montanide ISA-51 will be tested in ten patients with metastatic solid tumors. Patients will be treated with an ARG1 vaccine every third week for 45 weeks.

DETAILED DESCRIPTION:
Arginase-1 (ARG1) is an enzyme that converts the amino acid arginine into urea and ornithine. ARG1 is mainly expressed in hepatocytes but different myeloid cells are also capable of ARG1-expression.

An ARG1-induced arginine depletion suppresses T cell function through the impairment of the T cell receptor (TCR)-complex. A research group from the Center for Cancer Immune Therapy (CCIT) have identified spontaneous T cell reactivity against ARG1 peptides in peripheral blood mononuclear cells of cancer patients and healthy donors. The theoretic background for an ARG1 peptide vaccine is to activate ARG1-specific T cells to infiltrate the tumor microenvironment and eliminate ARG1-expressing immunosuppressive cells. The aim is to treat 10 patients with progressive solid tumors following treatment with standard of care agents. Patients will receive ARG1 vaccinations administered subcutaneously every third week for 45 weeks.

The primary endpoint is to evaluate safety and toxicity. Immune responses will be assessed using blood- and tumor tissue samples and clinical responses are evaluated using RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. The patient has metastatic solid tumors (NSCLC, colorectal cancer, urothelial cancer, breast cancer, ovarian cancer, malignant melanoma or HNSCC); progressive or recurrent disease on or following treatment with standard of care agents
3. At least one measurable parameter according to RECIST 1.1.
4. The patient has an ECOG performance status of 0 or 1
5. Life expectancy of at least 3 months
6. Prior PD1/PD-L1 allowed
7. The patient is a female of childbearing potential with negative pregnancy test
8. For fertile women: Agreement to use contraceptive methods with a failure rate of < 1 % per year during the treatment period and for at least 150 days 12 weeks after the treatment. Safe contraceptive methods for women are birth control pills, intrauterine device, contraceptive injection, contraceptive implant, contraceptive patch or contraceptive vaginal ring.
9. For men: Agreement to use contraceptive measures and agreement to refrain from donating sperm
10. The patient has met the following hematological and biochemical criteria:

    1. AST and ALT ≤2,5 X ULN or ≤5 X ULN with liver metastases
    2. Serum total bilirubin ≤1,5 X ULN or direct bilirubin ≤ ULN for patient with total bilirubin level > 1,5 ULN
    3. Serum creatinine ≤1,5 X ULN
    4. ANC (Absolute Neutrophil Count) ≥1,000/mcL
    5. Platelets ≥ 75,000 /mcL
    6. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
11. Mandatory provision of archival tissue and blood for biomarker testing at baseline
12. Mandatory provision of blood for biomarker testing during the study
13. Signed declaration of consent after oral and written information about the protocol

Exclusion Criteria:

1. The patient has not recovered from surgery or is less than 4 weeks from major surgery
2. The patient has a history of life-threatening or severe immune related adverse events on treatment with another immunotherapy and is considered to be at risk of not recovering
3. The patient is expected to require any other form of systemic antineoplastic therapy or radiation therapy while receiving the treatment. However, radiation therapy treatment of non target lesion is allowed.
4. The patient has a history of severe clinical autoimmune disease
5. The patient has a history of pneumonitis, organ transplant, human immunodeficiency virus positive, active hepatitis B or hepatitis C
6. The patient requires systemic steroids for management of immune-related adverse events experienced on another immunotherapy
7. The patient has any condition that will interfere with patient compliance or safety (including but not limited to psychiatric or substance abuse disorders)
8. The patient is pregnant or breastfeeding
9. The patient is unable to voluntarily agree to participate by signed informed consent or assent
10. The patient has an active infection requiring systemic therapy
11. The patient has received a live virus vaccine within 30 days of planned start of therapy
12. Significant medical disorder according to investigator; e.g. severe asthma or chronic obstructive lung disease, dysregulated heart disease or dysregulated diabetes mellitus
13. Concurrent treatment with other experimental drugs
14. Concurrent treatment with Valproate or Xanthin Oxidase inhibitors
15. Known side effects to Montanide ISA-51
16. Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
17. Severe allergy or anaphylactic reactions earlier in life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., MD, Study Director — CCIT-DK
Locations (1):
- Center for Cancer Immune Therapy Dept. of Hematology/oncology, Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorentzen CL, Martinenaite E, Kjeldsen JW, Holmstroem RB, Mork SK, Pedersen AW, Ehrnrooth E, Andersen MH, Svane IM. Arginase-1 targeting peptide vaccine in patients with metastatic solid tumors - A phase I trial. Front Immunol. 2022 Oct 17;13:1023023. doi: 10.3389/fimmu.2022.1023023. eCollection 2022. PMID 36330525

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARG1-18,19,20 Peptide Vaccine
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | ARG1-18,19,20 Peptide Vaccine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Median (Standard Deviation); unit: years] | 66 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 10

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Evaluated by CTCAE 4.0
Description: Patients were evaluated according to Common Terminology Criteria for Adverse Events (CTCEA). An adverse event (AE) is an abnormal clinical finding. Each participant was assessed from start of treatment until 6 months after the last vaccine.
Time Frame: 0 - 75 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ARG1-18,19,20 Peptide Vaccine
Number analyzed (Participants) | 10
Participants
  patients with worst AE grade 1 | 1
  patients with worst AE grade 2 | 7
  patients with worst AE grade 3 | 2
  patients with worst AE grade 4 | 0

2. Secondary Outcome: Immune Responses
Description: To evaluate the immunological impact of the ARG1-18,19,20 peptide vaccines using blood samples and tumor biopsies.
Time Frame: project blood samples were taken at baseline and every 3 months for a maximum of 1,5 year. Tumor biopsies were taken at baseline and after 3 months if possible.
Population: Development of a reactive T cell response against at least one of the ARG1 peptides during treatment using interferon-gamma ELISPOT
Measure: Count of Participants; unit: Participants
Arm/Group | ARG1-18,19,20 Peptide Vaccine
Number analyzed (Participants) | 10
Participants | 5

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) defined as time from treatment initiation to death, will be described with use of Kaplan Meier curve.
Time Frame: 0 - 75 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ARG1-18,19,20 Peptide Vaccine
Number analyzed (Participants) | 10
months | 7.3 [4.5 to 18.8]

4. Secondary Outcome: 4.Progression Free Survival
Description: Progression free survival (PFS) defined as the time from treatment initiation to disease progression, relapse or death due to any cause, which ever comes first, will be described with Kaplan Meier curve.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 0 - 75 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ARG1-18,19,20 Peptide Vaccine
Number analyzed (Participants) | 10
days | 62 [34.7 to 85.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at baseline and every 3 weeks (when the vaccine was given) for up to 6 months after the last vaccine ( 6 months follow-up)
Arm/Group | ARG1-18,19,20 Peptide Vaccine
All-Cause Mortality (participants affected / at risk) | 9/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARG1-18,19,20 Peptide Vaccine (N=10)
Ascites (Gastrointestinal disorders) | 1 — not related to study drug
Abdominal pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — not related to study drug
Facial paralysis (Nervous system disorders) | 1 — not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARG1-18,19,20 Peptide Vaccine (N=10)
Fatique (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Nausea (Gastrointestinal disorders) | 4
Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Dizziness (Nervous system disorders) | 3
Xerostomia (Gastrointestinal disorders) | 1
Granuloma at injection site (Skin and subcutaneous tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Mucositis (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Neuropathy (Nervous system disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Hypothyroidsm (Endocrine disorders) | 2
Transaminase elevation (Gastrointestinal disorders) | 7 — Only grade 1-2. Six of the seven patients had an increase in transaminases during treatment, however, they all had corresponding progression of metastatic lesion in the liver.
Anemia (Blood and lymphatic system disorders) | 3
Alkaline phosphate increased (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03689192/Prot_SAP_000.pdf